CLINICAL TRIAL: NCT01822054
Title: Childhood Body Composition and Brain Structure and Function
Status: Completed | Type: Observational
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 133540
Record Dates: First submitted 2013-02-26; First posted 2013-04-02 (Estimated); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Normal weight
- Obese

SUMMARY:
The specific aim of this research project is to use MRI methods to evaluate and compare brain structure and function in normal weight and obese children age 8-10 years.

ELIGIBILITY:
Inclusion Criteria:

* Healthy normal weight or obese children
* Parental report of full-term gestation
* Parental report of birth weight between 5th-95th percentiles
* Parental report of breastfeeding or cow's milk formula fed during infancy
* Right hand dominance

Exclusion Criteria:

* Maternal diabetes
* Maternal alcohol, tobacco or drug use during pregnancy
* Chronic sleep disorder
* History of psychological or psychiatric diagnosis
* History of neurological impairment or injury
* Surgical implant or other foreign object in the body which may be a MRI safety concern
* Dental work which may cause artifacts in MRI
* Claustrophobia
* High likelihood of inability to tolerate loud noise from the MRI scanner

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy normal weight or obese children (age 8-10 years)
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2012-01; Primary Completion 2013-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Brain structure | 8 - 10 years of age
  We will use high resolution volumetric MRI and DTIto measure the brain structure of these children

SECONDARY OUTCOMES:
Brain Function | 8-10 years of age
  We will use high resolution fMRI to measure the brain function under different cognitive paradigms

CONTACTS AND LOCATIONS:
Overall Officials: Xiawei Ou, PhD, Principal Investigator — Arkansas Children's Nutrition Center
Locations (1):
- Arkansas Children's Nutrition Center, Little Rock, Arkansas, United States